CLINICAL TRIAL: NCT06557577
Title: Evaluation of Hip Muscle Strength: Utility of an Adductor Fatigue Test to Substitute Handheld Dynamometry
Brief Title: Comparing an Adductor Fatigue Strength Test with Handheld Dynamometry
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Hugo Olmedillas Fernandez, Principal Investigator, University of Oviedo
Other Study IDs: UO2024/01
Record Dates: First submitted 2024-08-03; First posted 2024-08-16 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Groin Injury; Groin Strain
Keywords: Injury prevention; Strength assessment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy athletes: Competitive athletes without any groin injury.
  Interventions: Other: No intervention group.

INTERVENTIONS:
Other: No intervention group. — There is no intervention group.

SUMMARY:
The strength of the adductor muscles in a population of federated athletes will be measured using two tests: First, the maximum strength test, utilizing handheld dynamometry. Subsequently, endurance strength will be measured with the Adductor Fatigue Test (Brazilian Adductor Performance Test), in order to evaluate a possible correlation between the two tests.

DETAILED DESCRIPTION:
The strength of the adductor muscles in a population of federated athletes will be measured using two tests: First, the maximum strength test, utilizing dynamometry, where the subject will perform a maximal isometric contraction against the resistance provided by the investigator. Subsequently, endurance strength will be measured with the Adductor Fatigue Test (Brazilian Adductor Performance Test), the participant must perform an adductor exercise as many repetitions as possible until exhaution. In order to evaluate a possible correlation between the two tests and thus, by performing one of them, obtain the results of the other variable.

Apart from the strength measurements, democraphic caracteristics will be recorded to assess possible correlations between studied variables.

ELIGIBILITY:
Inclusion Criteria:

* Having an active lifestyle
* Competing at any level in a federated sports discipline.

Exclusion Criteria:

* Not consenting to participate in the research.
* Being unable to understand or write in Spanish.
* Having sustained any type of injury to the inguinal musculature in the past 3 months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Competitive athletes without groin injury in the last 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Maximal adductor strength | September to December (2024)
  Measuring the maximum strength of the adductor musculature, performed manually by a physiotherapist using a dynamometer over a brief working period. To begin the test, the subject should lie in a supine position on a flat surface. Their hip should be positioned at a 0º angle in our case. Ideally, at least three measurements should be taken, including a brief rest (~30 seconds) between each repetition to minimize muscle fatigue.
  The dynamometer should be placed between both ankles of the patient, with the forearm of the analyzing physiotherapist positioned in the middle as resistance. The patient should exert as much pressure as possible against the dynamometer, which is held by the physiotherapist, and against the physiotherapist's elbow, as if trying to close their legs like scissors, using their adductor muscles and maintaining the contraction for 5 seconds.
Adductor fatigue strength test | September to December (2024)
  The individual will begin by assuming a side plank position, supported by the elbow, bent, and the forearm (lower arm) on the ground. The hand of the supporting arm is placed on the waist of the side of the lower limb that is to be evaluated (the highest). The evaluated limb is supported by a 0.5-meter high bench at the ankle region, while the opposite limb does not touch the ground, remaining in a semi-flexed position. The subject must control the descent of the pelvis by performing a hip abduction until the pelvis lightly touches the ground, and then return to the initial position by raising the pelvis again. The score is defined as the maximum number of repetitions completed before reaching muscle failure. During the test, participants are instructed to keep both legs parallel and to ensure that the knee of the non-evaluated leg remains in a semi-flexed position. Maintaining the correct alignment of the trunk throughout the exercise is crucial.

SECONDARY OUTCOMES:
Weight | September to December (2024)
  Weight (kg)
Hip and groin outcome score (HAGOS) | September to December (2024)
  A questionnaire will be given to every participant to obtain information on groin pain symptoms in the last week. Minimum: 0; Maximum: 100. Higher scores mean better hip and groin health.
Age | September to December (2024)
  Age (in years)
Sex | September to December (2024)
  Biological sex
Leg length | September to December (2024)
  Leg length (in cm from the anterior superior iliac spine to the medial malleoulus)
Height | September to December (2024)
  Height (in cm)
Previous groin injury. | September to December (2024)
  Previous groin injury (in the last 3 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Escuela Profesional de Medicina de la Educación Fisica y el Deporte, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Queiroz JHM, Frota JP, Dos Reis FA, de Oliveira RR. Development and Predictive Validation of the Brazilian Adductor Performance Test for Estimating the Chance of Hip Adductor Injuries in Elite Soccer Athletes. Int J Sports Physiol Perform. 2023 Apr 20;18(6):653-659. doi: 10.1123/ijspp.2022-0306. Print 2023 Jun 1. PMID 37080542
- [Background] Robaina BQ, Medeiros DM, Roberti LS, Franke RA, Baroni BM. The Single Leg Bridge Test does not replace handheld dynamometer hamstring tests in a clinical setting. Phys Ther Sport. 2023 Sep;63:126-131. doi: 10.1016/j.ptsp.2023.08.001. Epub 2023 Aug 6. PMID 37573852